CLINICAL TRIAL: NCT05234996
Title: The Immersive Experience of Virtual Reality During Chemotherapy in Patients With Early Breast and Gynecological Cancers: the Patient's Dream Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, FABI ALESSANDRA, Principal Investigator, Regina Elena Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1105/18
Record Dates: First submitted 2021-12-31; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; virtual reality; supportive care
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality (Active Comparator): In The VRE arm, patients will use Virtual Reality headset (VR Headset), containing a selection of audiovisual productions made with 360 degrees technology and selected on the basis of content, plot and production dynamics. During the entire experience, an operator dedicated to patient care will be present to allow the most possible comfortable experience.
  Interventions: Device: 3 Virtual Reality headset (VR Headset),
- control arm (Active Comparator): In control arm, patients will entertain themselves with conventional means such as listening to music, watching a mobile program, reading newspapers, books, magazines or also doing nothing, according to the patient's preferences
  Interventions: Device: 3 Virtual Reality headset (VR Headset),

INTERVENTIONS:
Device: 3 Virtual Reality headset (VR Headset), — The VRE will administer through the use of 3 Virtual Reality headset (VR Headset), containing a selection of audiovisual productions made with 360 degrees technology and selected on the basis of content, plot and production dynamics.

SUMMARY:
"Patient's dream" study is a two-arm randomized controlled trial that will be conducted at Regina Elena National Cancer Institute, IRCCS (Rome), from April 2019 to January 2020. Before starting the first course of chemotherapy, patients will be randomly divided to receive the VRE (VRE arm) as "distraction therapy", or to entertain themselves with conventional means such as listening to music, watching a mobile program, reading newspapers, books, magazines or also doing nothing, according to the patient's preferences and for the entire duration of administration of the first CT cycle (control arm). A clinical team composed of three oncologists, three psychologists, one nurse and one expert VR operator will support the patients involved in the study.

The primary aims were the assessment of psychological distress, anxiety and quality of life between the two study arms. Secondary endpoints were the perceived time during the first course of CT and the acute and late toxicity.

The study will conduct in accordance with the ethical standards as laid down in the Declaration of Helsinki and its later amendments and within the protocol approved by the Central Ethics Committee (Trial registration number: RS 1105/18). A written informed consent will obtain from all participants included in the study.

ELIGIBILITY:
Inclusion Criteria

* diagnosis of breast or ovarian cancer confirmed histologically, from I to III stage;
* surgery as first therapeutic approach (in case of ovarian cancer, patients with minimal residual disease after surgery will be also included)
* first cycle of adjuvant CT, with or without a biological treatment according to the specific cancer (regimens including anthracyclines/taxanes, anthracyclines/cyclophosphamide, carboplatinum/taxane combined or not with trastuzumab for breast cancer, carboplatin/paclitaxel combined or not with bevacizumab for ovarian cancer);
* aged ≥ 18 years;
* performance status (ECOG) 0-2;
* life expectancy > 12 months;
* ability to understand and sign the informed consent.

Exclusion Criteria:

* presenting prior history of seizures;
* disorders of the mood;
* previous history of alcohol and/or drug addiction;
* disorder of vision and eyes;
* history of psychiatric pathologies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
evaluation of Distress | Questionnaire is administered during three times: at baseline, after the somministration of the first cycle of chemotherapy and after 21 days, before the start of the second cycle. Each cycle in 21 days
  Distress is evaluate with HAds questionnaire
evaluation of Quality of life | Questionnaire is administered during three times: at baseline, after the somministration of the first cycle of chemotherapy and after 21 days, before the start of the second cycle. Each cycle in 21 days
  Quality of life is evaluate with QLQ-C30- BR23

SECONDARY OUTCOMES:
Evaluation of Incidence of treatment-emergent adverse events | Questionnaire is administered during three times: at baseline, after the somministration of the first cycle of chemotherapy and after 21 days, before the start of the second cycle. Each cycle in 21 days
  this incidence in evaluate and classified with the Common Terminology Criteria for Adverse Events (CTCAE 5.0)
Evaluation of Patients Report Outcomes | Questionnaire is administered during three times: at baseline, after the somministration of the first cycle of chemotherapy and after 21 days, before the start of the second cycle. Each cycle in 21 days
  This outcomes is evaluated with PROs

CONTACTS AND LOCATIONS:
Overall Officials: Fabi Alessandra, Study Director — Regina Elena Cancer Institute
Locations (1):
- alessandra Fabi, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fabi A, Fotia L, Giuseppini F, Gaeta A, Falcicchio C, Giuliani G, Savarese A, Taraborelli E, Rossi V, Malaguti P, Giannarelli D, Pugliese P, Cognetti F. The immersive experience of virtual reality during chemotherapy in patients with early breast and ovarian cancers: The patient's dream study. Front Oncol. 2022 Sep 30;12:960387. doi: 10.3389/fonc.2022.960387. eCollection 2022. PMID 36249001